CLINICAL TRIAL: NCT07399522
Title: A Randomized Controlled Trial of Home-Based Calligraphic Handwriting Exercises in Patients With Parkinson's Disease
Brief Title: Home-Based Calligraphic Handwriting Exercises in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Llamas Velasco (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor-Investigator, Sara Llamas Velasco, Postdoctoral Researcher in Neurology, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI21-01622
Record Dates: First submitted 2026-01-21; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: PARKINSON DISEASE (Disorder)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calligraphic Handwriting Exercise Program (Experimental): Participants assigned to this group will perform a structured home-based calligraphic handwriting exercise program designed to improve fine motor control and manual dexterity over a 12-week period.
  Interventions: Behavioral: Calligraphic Handwriting Exercise Program
- Usual Care (No Intervention): Participants assigned to this group will receive usual clinical care and will not participate in the calligraphic handwriting exercise program during the study period.

INTERVENTIONS:
Behavioral: Calligraphic Handwriting Exercise Program — A structured home-based calligraphic handwriting exercise program designed to train fine motor control and manual dexterity. Participants perform predefined handwriting exercises regularly over a 12-week period using provided written materials.
  Arms: Calligraphic Handwriting Exercise Program

SUMMARY:
Parkinson's disease is a progressive neurodegenerative disorder with no curative treatment currently available. Its symptoms lead to increasing limitations in daily activities, with impairments in manual dexterity being particularly relevant. Handwriting difficulties are common in patients with Parkinson's disease; however, it remains unclear whether a rehabilitation program based on handwriting exercises can improve overall manual dexterity and daily functioning.

This randomized, single-blind controlled trial aims to evaluate the effects of a 12-week home-based calligraphic handwriting exercise program on manual dexterity in patients with Parkinson's disease. Participants will be recruited from the Movement Disorders Clinic of Hospital 12 de Octubre (Madrid, Spain) and randomly assigned to either an intervention group or a control group.

Manual dexterity will be primarily assessed using the Purdue Pegboard Test across scheduled study visits. Secondary outcomes will include measures of dexterity related to activities of daily living, quality of life, and motor function.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients aged 40 to 80 years
* Clinical diagnosis of Parkinson's disease according to the UK Brain Bank criteria.
* Hoehn and Yahr stage 1 to 4
* Assessed in the ON-medication state (approximately 90 minutes after levodopa intake)
* Stable antiparkinsonian treatment for at least 4 weeks prior to study entry and maintained throughout the study period

EXCLUSION CRITERIA:

* Parkinson's disease-related dementia, defined as a Montreal Cognitive Assessment (MoCA) score < 21
* Upper limb comorbidities unrelated to Parkinson's disease that could interfere ith exercise performance (e.g., arthritis, recent fractures, stroke sequelae, or peripheral neuropathy)
* Severe tremor or severe dyskinesias affecting the dominant hand, defined as:

  * a score ≥ 3 on UPDRS-III items 20 or 22, or
  * score ≥ 2 on UPDRS-IV item 33

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Change in Manual Dexterity | Baseline and up to 12 weeks
  Manual dexterity will be assessed using the Purdue Pegboard Test. The primary outcome will be the change in Purdue Pegboard Test score from baseline across scheduled study visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No